CLINICAL TRIAL: NCT03039868
Title: Use of Pap Smear Derived Cells to Analyze the Expression of SLC6A14 and GPR81 Genes
Status: Terminated | Type: Observational
Why Stopped: results were not as hypothesized
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Other Study IDs: L17-030
Record Dates: First submitted 2017-01-30; First posted 2017-02-01 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — RNA will be extracted from Pap smear cells for further analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal Pap smears: This is the control group.
- Abnormal Pap smears: This is the case group.

SUMMARY:
SLC6A14 may serve as a biomarker for cervical dysplasia or cervical cancer.

DETAILED DESCRIPTION:
SLC6A14 amino acid transporter Previous research has shown that the expression of the amino acid transporter SLC6A14 is up-regulated in cervical cancer1. Studies on breast, colon and pancreatic cancer cells have shown that SLC6A14 amino acid transporter serves the role of supporting amino acid nutrition to these cancer cells2,3,4. It has also been shown that genetic deletion or pharmacologic blockade of the above transporter will suppress the growth of the tumor cells both in vitro and in vivo4,5,6.

We are interested in exploring the expression of SLC6A14 transporter in normal cervical epithelial cells, in cervical dysplasia and cervical cancer; and to see if expression of this transporter has any correlation to presence/severity of cervical dysplasia/cancer, and also to see if this may serve as a biomarker to predict or diagnose the presence of cervical dysplasia and cervical cancer.

GPR81, a G-protein coupled receptor for lactate Human vagina is predominantly colonized by Lactobacilli, which convert glycogen in the vaginal epithelial cells to lactic acid. Some species of Lactobacilli also produce hydrogen peroxide. Both lactate and H2O2 help to keep the vaginal pH low (acidic <4.5) and also help in preventing colonization of the vagina by pathogenic bacteria. When the levels of Lactobacilli in the vaginal micro environment change (as with certain vaginal infections, decline in estrogen levels etc), levels of lactate decline and H2O2 decline-thus predisposing women to vaginal infections.

Vaginal and cervical fluids contain lactate in millimolar concentrations. Recent studies have identified a G-protein-coupled cell-surface receptor for lactate,-called GPR81. Studies from Dr. Ganapathy's lab have shown that activation of the receptor GPR81 in B lymphocytes enhances the production of IgA antibody, which plays a role in defense mechanisms of mucosal surfaces. IgA antibodies are seen in high levels in the intestinal, colonic, lung mucosa as well as vaginal epithelial surfaces. These IgA antibodies protect the colonization of mucosal surfaces by pathogenic bacteria. Thus GPR 81 is an anti-inflammatory molecule. Hence it may inversely correlate with cervical dysplasia. We propose to investigate if the vaginal and cervical epithelial cells express this GPR81, whether GPR81 expression correlates to cervical dysplasia.

If a correlation exists between lactate levels and GPR81 expression, declining Lactobacilli levels with associated decline in lactate levels, could lead to decreased GPR81 expression on epithelial cells, and thus decline in IgA antibody secretion. This could be the reason for vaginal infections with decreased Lactobacilli. If infection with HPV virus occurs, this will lead to abnormalities in the Pap smear and potential cervical dysplasia in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Women who present to the TTUHSC Lubbock OBGYN Clinics for exams and are having cervical Pap smear collected as part of the evaluations.
2. Women who have vaginal discharge will be also included in the study if they are having cervical Pap smear collected as part of their exam.
3. Age criteria 21yr- 65yrs or more -per ASCCP guidelines for Pap smears.
4. Patients on any medications will also be included- medications have no effect on Pap smear results.

Exclusion Criteria:

1. Women who have had a hysterectomy.
2. Women having vaginal Pap smears.
3. Women with known HIV.

Ages: 21 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll a minimum of 150 and a maximum of 400 subjects. The subjects will all be women who present to the Texas Tech Obstetrics and Gynecology Clinics for exams and are having cervical Pap smear collected as part of their exams. The study subjects will be recruited after informed consent is obtained and they agree to the collection of 1-2 additional cervical Pap smear specimens to be used for the research study.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Expression of SLC6A14 and GPR81 transporter in cervical epithelial cells measured as "delta Ct" to correlate expression levels to cervical dysplasia and cervical cancer | Prospective study over a period of 3 years.

IPD SHARING:
Plan to Share IPD: No